CLINICAL TRIAL: NCT02240875
Title: A Phase Ia, Dose-Escalating, Safety and Immunogenicity Trial of the Monovalent Zaire Ebola Viral Vector Candidate Vaccine cAd3-EBO Z and the Heterologous Prime-boost Candidate Vaccine Regimen cAd3-EBO Z and MVA-BN® Filo in Healthy UK Adults
Brief Title: A Study to Assess New Ebola Vaccines, cAd3-EBO Z and MVA-BN® Filo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBL01; 2014-003518-10 (EudraCT Number)
Record Dates: First submitted 2014-09-10; First posted 2014-09-16 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Ebola; Ebola Zaire
Keywords: Ebola; Zaire
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Group 1 (Experimental): Single dose of cAd3-EBO Z at 1 x 10^10 vp intramuscularly
  Interventions: Biological: cAd3-EBO Z at 1 x 10^10 vp
- Group 1b (Experimental): Single dose of cAd3-EBO Z at 1 x 10^10 vp intramuscularly, followed by 4.4x10^8 TCID50s MVA-BN® Filo
  Interventions: Biological: cAd3-EBO Z at 1 x 10^10 vp; Biological: 4.4x10^8 TCID50s MVA-BN® Filo
- Group 1c (Experimental): Single dose of cAd3-EBO Z at 1 x 10^10 vp intramuscularly, followed by 2.2x10^8 TCID50s MVA-BN® Filo
  Interventions: Biological: cAd3-EBO Z at 1 x 10^10 vp; Biological: 2.2x10^8 TCID50s MVA-BN® Filo
- Group 2 (Experimental): Single dose of cAd3-EBO Z at 2.5 x 10^10 vp intramuscularly
  Interventions: Biological: cAd3-EBO Z at 2.5 x 10^10 vp
- Group 2b (Experimental): Single dose of cAd3-EBO Z at 2.5 x 10^10 vp intramuscularly, followed by 4.4x10^8 TCID50s MVA-BN® Filo
  Interventions: Biological: cAd3-EBO Z at 2.5 x 10^10 vp; Biological: 4.4x10^8 TCID50s MVA-BN® Filo
- Group 2c (Experimental): Single dose of cAd3-EBO Z at 2.5 x 10^10 vp intramuscularly, followed by 2.2x10^8 TCID50s MVA-BN® Filo
  Interventions: Biological: cAd3-EBO Z at 2.5 x 10^10 vp; Biological: 2.2x10^8 TCID50s MVA-BN® Filo
- Group 3 (Experimental): Single dose of cAd3-EBO Z at 5 x 10^10 vp intramuscularly
  Interventions: Biological: cAd3-EBO Z at 5 x 10^10 vp
- Group 3b (Experimental): Single dose of cAd3-EBO Z at 5 x 10^10 vp intramuscularly, followed by 4.4x10^8 TCID50s MVA-BN® Filo
  Interventions: Biological: cAd3-EBO Z at 5 x 10^10 vp; Biological: 4.4x10^8 TCID50s MVA-BN® Filo
- Group 3c (Experimental): Single dose of cAd3-EBO Z at 5 x 10^10 vp intramuscularly, followed by 2.2x10^8 TCID50s MVA-BN® Filo
  Interventions: Biological: cAd3-EBO Z at 5 x 10^10 vp; Biological: 2.2x10^8 TCID50s MVA-BN® Filo
- Group 4 (Experimental): Single dose of cAd3-EBO Z at 2.5 x 10^10 vp intramuscularly at day 0, followed by 2.2 x 10^8 TCID50s MVA-BN® Filo at day 7
  Interventions: Biological: cAd3-EBO Z at 2.5 x 10^10 vp; Biological: 2.2x10^8 TCID50s MVA-BN® Filo
- Group 5 (Experimental): Single dose of cAd3-EBO Z at 2.5 x 10^10 vp intramuscularly at day 0, followed by 2.2 x 10^8 TCID50s MVA-BN® Filo at day 14
  Interventions: Biological: cAd3-EBO Z at 2.5 x 10^10 vp; Biological: 2.2x10^8 TCID50s MVA-BN® Filo
- Group 6 (Experimental): Single dose of cAd3-EBO Z at 2.5 x 10^10 vp intramuscularly at day 0, followed by 4.4 x 10^7 TCID50s MVA-BN® Filo at day 7
  Interventions: Biological: cAd3-EBO Z at 2.5 x 10^10 vp; Biological: 4.4 x 10^7 TCID50s MVA-BN® Filo
- Group 7 (Experimental): Single dose of cAd3-EBO Z at 2.5 x 10^10 vp intramuscularly at day 0, followed by 4.4 x 10^7 TCID50s MVA-BN® Filo at day 14
  Interventions: Biological: cAd3-EBO Z at 2.5 x 10^10 vp; Biological: 4.4 x 10^7 TCID50s MVA-BN® Filo

INTERVENTIONS:
Biological: cAd3-EBO Z at 1 x 10^10 vp — Low dose cAd3-EBO Z
  Arms: Group 1; Group 1b; Group 1c
Biological: cAd3-EBO Z at 2.5 x 10^10 vp — Medium dose cAd3-EBO Z
  Arms: Group 2; Group 2b; Group 2c; Group 4; Group 5; Group 6; Group 7
Biological: cAd3-EBO Z at 5 x 10^10 vp — High dose cAd3-EBO Z
  Arms: Group 3; Group 3b; Group 3c
Biological: 4.4x10^8 TCID50s MVA-BN® Filo — High dose MVA-BN® Filo
  Arms: Group 1b; Group 2b; Group 3b
Biological: 2.2x10^8 TCID50s MVA-BN® Filo — Low dose MVA-BN® Filo
  Arms: Group 1c; Group 2c; Group 3c; Group 4; Group 5
Biological: 4.4 x 10^7 TCID50s MVA-BN® Filo — Very low dose MVA-BN® Filo
  Arms: Group 6; Group 7

SUMMARY:
The purpose of this study is to assess two new Ebola vaccines: cAd3-EBO Z at 3 different doses, and a second vaccine, MVA-BN® Filo, at 3 different doses. The study will enable us to assess the safety of the vaccines and the extent of the immune response in healthy volunteers. The investigators will do this by giving volunteers a either one or two vaccinations, doing blood and saliva tests and collecting information about any symptoms that occur after vaccination. This is the first trial to use either of these vaccines in humans. We plan to recruit a total of 92 volunteers to be vaccinated.

DETAILED DESCRIPTION:
Long- term immunology follow-up: In order to assess the durability of vaccine induced immunogenicity, all vaccinated subjects will be invited back to attend a maximum of 3 further optional follow up visits at least 12 months after their final vaccination. The 3 visits will have a minimum interval of 3 months between them, and the final visit must take place no longer than 12 months after the first optional visit.

Volunteers who attend these visits will be asked about occurrence of any SAEs during the intervening period. SAE data for this period will not be collected in those volunteers who decline to attend these additional visits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their general practitioner (GP)
* For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational Ebola or Marburg vaccine, a chimpanzee adenovirus vectored vaccine or any other investigational vaccine likely to impact on interpretation of the trial data
* Receipt of any live, attenuated vaccine within 28 days prior to enrolment
* Receipt of any subunit or killed vaccine within 14 days prior to enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, (e.g. egg products) including urticaria, respiratory difficulty or abdominal pain
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Poorly controlled asthma or thyroid disease
* Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venepuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Current anti-tuberculosis prophylaxis or therapy
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Travel to a Ebola or Marburg endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis (see Appendix A and Appendix B)
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the Ebola Zaire vaccine cAd3-EBO Z when administered to healthy volunteers at 3 doses | 6 months
  The specific endpoints for safety and reactogenicity will be actively and passively collected data on adverse events.

SECONDARY OUTCOMES:
Cellular and humoral immunogenicity of the Ebola Zaire vaccine cAd3-EBO Z when administered to healthy volunteers at 3 doses | 6 months
  The primary immunogenicity outcome measures are ELISA and neutralization antigen-specific assays for antibody responses and intracellular cytokine staining (ICS) assay for T cell responses.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian V Hill, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Lambe T, Rampling T, Samuel D, Bowyer G, Ewer KJ, Venkatraman N, Edmans M, Dicks S, Hill AV, Tedder RS, Gilbert SC. Detection of Vaccine-Induced Antibodies to Ebola Virus in Oral Fluid. Open Forum Infect Dis. 2016 Feb 22;3(1):ofw031. doi: 10.1093/ofid/ofw031. eCollection 2016 Jan. PMID 27004234
- [Derived] Ewer K, Rampling T, Venkatraman N, Bowyer G, Wright D, Lambe T, Imoukhuede EB, Payne R, Fehling SK, Strecker T, Biedenkopf N, Krahling V, Tully CM, Edwards NJ, Bentley EM, Samuel D, Labbe G, Jin J, Gibani M, Minhinnick A, Wilkie M, Poulton I, Lella N, Roberts R, Hartnell F, Bliss C, Sierra-Davidson K, Powlson J, Berrie E, Tedder R, Roman F, De Ryck I, Nicosia A, Sullivan NJ, Stanley DA, Mbaya OT, Ledgerwood JE, Schwartz RM, Siani L, Colloca S, Folgori A, Di Marco S, Cortese R, Wright E, Becker S, Graham BS, Koup RA, Levine MM, Volkmann A, Chaplin P, Pollard AJ, Draper SJ, Ballou WR, Lawrie A, Gilbert SC, Hill AV. A Monovalent Chimpanzee Adenovirus Ebola Vaccine Boosted with MVA. N Engl J Med. 2016 Apr 28;374(17):1635-46. doi: 10.1056/NEJMoa1411627. Epub 2015 Jan 28. PMID 25629663